CLINICAL TRIAL: NCT01108016
Title: Expanding Rural Access: Distance Delivery of Support Groups (Main Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Cheryl Koopman, Stanford University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SU-03012010-5082; BRSADJ0019
Record Dates: First submitted 2010-04-14; First posted 2010-04-21 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Depression; Breast Cancer; Stress; Breast Cancer Non-invasive Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer Metastatic Breast Cancer
MeSH Terms: conditions — Depression; Breast Neoplasms

INTERVENTIONS:
Behavioral: Videoconferencing support group

SUMMARY:
The study will answer two questions about women with breast cancer in rural communities:

1. Will they find this support group format utilizing videoconferencing acceptable and rewarding?
2. Will they report a greater sense of emotional and informational support, and less depression and traumatic stress, than the control groups of women who wait to participate until after the first groups have ended?

ELIGIBILITY:
Inclusion Criteria:To be eligible to participate, a woman must meet all of the following criteria:

1. be a resident of one of nine rural counties in northeastern California (Modoc, Plumas, Siskiyou, Shasta, Lassen, Trinity, Sierra, Nevada, and Tehama),
2. be able to travel to a rural health facility included in the Northern Sierra Rural Health Network to participate in videoconferencing meetings;
3. be able to speak and read English well enough to be able to read, discuss, and comprehend the consent form;
4. be 21 years of age or older;
5. have been diagnosed with breast cancer by a physician; and
6. who (in the judgment of the Local Coordinator) is not unduly distressed or otherwise not able to participate effectively in a support group.

Women will be included with any stage of breast cancer as our pilot study demonstrated that in these rural communities, women wanted to include women with any stage of breast cancer in their groups. Also, our pilot study results showed that it worked fine to include women regardless of the period elapsing since they received their diagnosis, as our pilot study results showed that some women with a long period of time elapsing since receiving their diagnosis were still in need of a source of social support for coping with having had this experience and felt that they had a lot of help to offer women who had more recently received a breast cancer diagnosis. The 9 counties were selected because they are among the most remote counties in California, yet they have strong primary care systems in place, and most patients receive specialty care in-state, as opposed to out-of-state. Every effort will be made to include women of ethnic minority groups.

The support group facilitator, community advisory board (CAB) members, and the local community coordinators will also be recruited for the interviews, with informed consent, identified by having played one of these roles for this study.

Exclusion Criteria:Potential participants who do not meet all of the inclusion criteria listed above will be excluded.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Intensity and frequency of posttraumatic stress symptoms in the past month as assessed by total score on the Posttraumatic Check List - Specific version (PCL-S) for breast cancer. | after 8 weeks of the immediate group sessions
Intensity and frequency of depression symptoms in the past week as assessed by total score on the Center for Epidemiological Studies Depression scale (CES-D) | after 8 weeks of the immediate group sessions

SECONDARY OUTCOMES:
Intensity and frequency of emotional control as assessed by the total score on the Courtauld Emotional Control Scale (CECS), | after 8 weeks of the immediate group sessions
Level of self-efficacy for coping with breast cancer as assessed by the total score on the Cancer Behavior Inventory (CBI). | after 8 weeks of the immediate group sessions
Satisfaction with social support as assessed by the total satisfaction score on the UCLA Social Support Inventory. | after 8 weeks of the immediate group sessions

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Koopman, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States